CLINICAL TRIAL: NCT06009861
Title: Neoadjuvant Chemoimmunotherapy With Tislelizumab, Albumin-bound Paclitaxel, and Cisplatin in Locally Advanced Oral/Oropharyngeal Squamous Cell Carcinoma: A Prospective, Multicenter, Single-arm Study
Brief Title: Neoadjuvant Tislelizumab Plus Chemotherapy for Locally Advanced Oral/Oropharyngeal Cancer (NeoSPOT)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Hospital of Stomatology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUSSIRB-202386047
Record Dates: First submitted 2023-08-16; First posted 2023-08-24 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Oral Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab; Albumin-Bound Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Tislelizumab plus chemotherapy and adjuvant RT or Tislelizumab plus CCRT (Experimental): Neoadjuvant phase: Patients will receive neoadjuvant Tislelizumab in combination with Albumin-Bound Paclitaxel and Cisplatin Q3W for 2 cycles.
  Adjuvant phase:
  For High-risk group(non-R0 resection or extranodal extension (ENE) or Lymph node metastasis>5): Concurrent chemoradiotherapy followed by Tislelizumab Q3W for 14 cycles.
  For the other group: intensity-modulated radiation therapy.
  Interventions: Drug: Tislelizumab; Drug: Albumin-Bound Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Tislelizumab — Dose: 200 mg Route: Intravenous infusion Frequency & treatment mode: Day 1, every 3 weeks
Drug: Albumin-Bound Paclitaxel — Dose: 260 mg/m^2 Route: Intravenous infusion Frequency & treatment mode: Day 1, every 3 weeks
Drug: Cisplatin — Dose: 60-75 mg/m^2 Route: Intravenous infusion Frequency & treatment mode: Day 1, every 3 weeks

SUMMARY:
Previous studies confirmed locally advanced oral/oropharyngeal squamous cell carcinoma (LA OSCC or OPSCC) patients with a pathological response had higher probability of survival in neoadjuvant settings. Several ongoing trials of neoadjuvant immunotherapy in head and neck cancer showed promising results. However, the optimal regimen remains unclear. This trial aimed to evaluate the efficacy and safety of neoadjuvant therapy with anti-programmed cell death 1 monoclonal antibody Tislelizumab and chemotherapy, followed by surgery and adjuvant radiotherapy or chemoradiotherapy plus Tislelizumab in LA OSCC or OPSCC.

ELIGIBILITY:
Inclusion Criteria:

* Cytological or histological diagnosis of initially or potentially surgically resectable Local advanced oral/oropharyngeal squamous cell carcinoma (stage III-IV).
* Plan to proceed neoadjuvant therapy.
* No prior anti-cancer treatment (include surgery, radiotherapy and systemic therapy) for oral/oropharyngeal squamous cell carcinoma.
* Clinically evaluable lesions per RECIST1.1.
* The age of signing the informed consent is 18-80 years old, regardless of gender.
* ECOG performance score 0-1.
* Estimated survival time≥6 months (this criterion overlaps with other inclusion criteria and must meet the following: ECOG score 0-1; Vital organ function meets the inclusion criteria in Article 8; Oral or oropharyngeal cancer does not involve the internal carotid artery; No subcutaneous metastases; No distant metastasis).
* Adequate organ function as follows: 1) Leukocyte count ≥ 3,000/mm3; 2) Absolute neutrophil count ≥ 1,500/mm3; 3) Platelet count ≥ 100,000/mm3; 4) Hemoglobin ≥ 90 g/L; 5) Serum creatinine ≤ 1.5 × ULN OR CrCl≥50 ml/min（Cockcroft-Gault）; 6) Total bilirubin ≤ 1.5 × upper limit of normal (ULN); 7) AST (SGOT) and ALT (SGPT) < 2.5 × ULN;
* Subjects able and willing to follow research and follow-up procedures.
* For male and female subjects of childbearing age must agree to use adequate contraception throughout the study period and for 6 months after the end of treatment.
* Subjects voluntarily joined the clinical study and signed the informed consent.

Exclusion Criteria:

* Previous therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 or any other antibody targeting T cell co-regulatory pathways.
* History of allergy, and may have a potential allergy or intolerance to the investigational drug and its similar biologics.
* Participated in clinical trials of other antitumor drugs within 4 weeks prior to initial administration; Or receive live attenuated vaccine within 4 weeks prior to initial administration or during the study period;
* Subjects with concurrent other active malignancies. History of other types for cancer within past 5 years (exclude adequately treated skin squamous cell carcinoma or controlled skin basal cell carcinoma).
* Advanced subjects with symptoms, visceral dissemination, and a short-term risk of life-threatening complications (including uncontrolled massive exudation [pleural, pericardial, peritoneal], pulmonary lymphangitis, and more than 30% liver involvement).
* Subjects with active autoimmune disease or history of refractory autoimmune disease.
* Subjects with grade II or higher myocardial ischemia or myocardial infarction, uncontrolled arrhythmia (including QTc interval ≥450 ms in men and ≥470 ms in women), NYHA class III-IV cardiac insufficiency, or left ventricular ejection fraction (LVEF) <50% on echocardiography, myocardial infarction within 6 months before enrollment, New York Heart Association class II or higher heart failure, uncontrolled angina, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease, or electrocardiogram suggestive of acute ischemia or active conduction system abnormalities;
* Severe infection (e.g. requiring intravenous antibiotics, antifungal or antiviral medication) within 4 weeks before first dose, or unexplained fever >38.5°C during screening/before first dose;
* Subjects with a history of abuse of psychotropic substances and unable to withdraw from them or with mental disorders;
* Subjects undergone major surgery or have an open wound or fracture within 4 weeks before the first dose;
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (positive hepatitis C antibody and HCV-RNA above the lower limit of detection of the analytical method) or co-infection of hepatitis B and hepatitis C;
* Central nervous system metastasis;
* Subjects with a history of genetic or acquired bleeding or coagulation dysfunction (eligibility criteria at the investigator's discretion);
* Other conditions that the investigator determined were inappropriate for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Event free survival (EFS) at 2 years | Up to 2 years
  EFS is the time from the date of randomization to the date of first record of any of the following events: disease progression; local or distant recurrence as assessed with imaging or biopsy as indicated; or death due to any cause.

SECONDARY OUTCOMES:
Major Pathological Response (mPR) | Up to 30 days post-surgery
  The proportion of participants with a major pathological response (mPR) as assessed by the Central Pathologist at the time of definitive surgery. mPR is defined as ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen and all the sampled regional lymph nodes.
Pathological Complete Response (pCR) | Up to 30 days post-surgery
  Pathological complete response (pCR) is measured as the proportion of participants with a pathological complete response as assessed by the central pathologist at the time of definitive surgery. pCR is defined as having no residual invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes.
Overall response rate (ORR) | UP to 30 days prior-surgery
  Overall response rate (ORR) is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria.
Overall survival (OS) | Up to 2 years
  OS is the time from randomization to death due to any cause.
Adverse events (AEs) | Up to 2 years
  Number of participants experiencing any sign, symptom, disease, or worsening of preexisting conditions temporally associated with the experimental interventions or irrespective of the experimental interventions per NCI-CTCAE V5.0.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Peking University School and Hospital Stomatology, Beijing, Beijing Municipality
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Affiliated Hospital of Chifeng College, Chifeng, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Hospital of Stomatology of Jilin University, Changchun, Jilin
  - China Medical University School and Hospital Of Stomatology, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No